CLINICAL TRIAL: NCT06706076
Title: A Phase 1/2 Open-Label, Multicenter, First-in-Human Study of the Safety, Tolerability, Pharmacokinetics, and Antitumor Activity of BH-30643 in Adult Subjects With Locally Advanced or Metastatic NSCLC Harboring EGFR and/or HER2 Mutations (SOLARA)
Brief Title: A Study of BH-30643 in Subjects With Locally Advanced or Metastatic NSCLC Harboring EGFR and/or HER2 Mutations
Acronym: SOLARA
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BlossomHill Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BH-30643-01
Record Dates: First submitted 2024-11-19; First posted 2024-11-26 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-11

CONDITIONS: NSCLC (Advanced Non-small Cell Lung Cancer)
Keywords: NSCLC; Locally Advanced NSCLC; Metastatic NSCLC; Non-small Cell Lung Cancer; HER2 mutation; EGFR mutation; EGFR classical mutation; EGFR atypical mutation; EGFR exon20 insertion; EGFR uncommon mutation; EGFR resistant mutation; BH-30643; Tyrosine kinase inhibitor; TKI; EGFR; OMNI-EGFR; EGFR kinase domain mutations; EGFR common mutation; EGFR activating mutation; Ex19del; EGFR del E746_A750; Exon 19 deletion; L858R; C797S; C797G; C797X; T790M; G719X; G724X; L718V; L718X; L861Q; S768I; S768X; E709X; L747X; Exon 19 insertion; L833X; L861X; V769X; V834X
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1 Dose Escalation and Expansion (Experimental): * BH-30643 monotherapy for dose escalation
  * BH-30643 monotherapy for dose expansion/optimization at doses determined from dose escalation data
  * BH-30643 twice daily oral dosing
  Interventions: Drug: BH-30643
- Phase 2 (Experimental): BH-30643 administered at the RP2D dose determined in Phase 1
  Interventions: Drug: BH-30643

INTERVENTIONS:
Drug: BH-30643 — BH-30643 will be provided as either 10 mg or 40 mg capsules. Subjects will take BH-30643 orally depending on their dose level assignment.
  Arms: Phase 1 Dose Escalation and Expansion
Drug: BH-30643 — BH-30643 will be provided as either 10 mg or 40 mg capsules. Subjects will take BH-30643 orally depending on their dose level assignment.
  Arms: Phase 2

SUMMARY:
This Phase1/2, open label, multicenter study will assess the safety, tolerability, pharmacokinetics (PK), pharmacodynamics and preliminary anti-tumor activity of BH-30643 in patients with NSCLC having EGFR and/or HER2 mutations.

Phase 1 will determine the recommended Phase 2 dose (RP2D) and, if applicable, the maximum tolerated dose (MTD) of BH-30643.

Phase 2 will further evaluate the antitumor efficacy and safety in specified cohorts determined by EGFR/HER2 mutation subtypes and/or treatment history at the RP2D, as well as the population PK.

DETAILED DESCRIPTION:
BH-30643 is a novel, orally available, non-covalent, macrocyclic, mutant selective OMNI-EGFR inhibitor that targets a broad diversity of mutations in the EGFR kinase domain. These include EGFR classical mutations (e.g., ex19del and L858R) as well as less common (atypical) mutations (including G719X, S768I, L861Q, E709X, and beyond). BH-30643 also overcomes a variety of mutations which can cause resistance to previously approved EGFR TKIs (including both C797S and T790M). BH-30643 was designed to be selective over wildtype EGFR and HER2.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years or legal adult.
* Pathologically confirmed diagnosis of locally advanced or metastatic NSCLC with EGFR (classical, atypical, exon20 insertion) or HER2 mutations in the kinase domain of exons 18, 19, 20, or 21. EGFR mutations include activating and acquired EGFR resistance mutations that might form compound mutations.
* Had received standard therapies.
* Has at least 1 measurable target extracranial lesion according to RECIST v1.1.
* Eastern Cooperative Oncology Group Performance Status ≤ 1.
* Has a life expectancy of ≥ 3 months.
* Has adequate hematologic, hepatic, and renal function. *The above are a summary; other Inclusion Criteria details may apply.

Exclusion Criteria:

* History of any concurrent malignancy within the previous 2 years.
* Known other oncogenic driver alterations (eg, moderate or high MET amplification) or histological transformation (eg, to small cell carcinoma, etc.).
* Unresolved toxicities from prior therapies.
* Any significant and uncontrolled medical condition, such as infection.
* History of interstitial lung disease from any cause
* Clinically significant cardiovascular event within 6 months or significant history of major organ.
* Actively receiving investigational therapy(ies) in another clinical study. *The above are a summary; other Exclusion Criteria details may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Estimated)
Dates: Start 2025-01-09 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLTs) (Phase 1, Dose Escalation) | Within the first 21 days of the first dose of BH-30643.
  Assess dose-limiting toxicities (DLTs) as defined in the study protocol.
Recommended Phase 2 dose (RP2D) (Phase 1, Dose Expansion/Optimization) | Within 21 days of last participant dosed during Dose Expansion/Optimization.
  Determine the RP2D for Phase 2.
Objective Response Rate (ORR) (Phase 2) | Approximately 3 years after the first participant dosed.
  Determine ORR as assessed by Blinded Independent Central Review (BICR).

SECONDARY OUTCOMES:
Safety | From enrollment through study completion, approximately 48 months.
  Assess incidence and severity of treatment-emergent adverse events (TEAEs), as defined by CTCAE, V5.0 (Phase 1 and Phase 2).
Area under the plasma concentration-time curve from time zero to time of the last quantifiable concentration (AUClast) of BH-30643 for Single dose (Phase 1). | Predose and up to 24 hours postdose.
  Determine area under the plasma concentration-time curve from time zero to time of the last quantifiable concentration (AUClast) of BH-30643.
Maximum observed plasma concentration (Cmax) of BH-30643 for Single dose (Phase 1). | Predose and up to 24 hours postdose.
  Determine maximum observed plasma concentration (Cmax) of BH-30643.
Time to reach Cmax (Tmax) of BH-30643 for Single dose (Phase 1). | Predose and up to 24 hours postdose.
  Determine time to reach Cmax (Tmax) of BH-30643.
Area under the plasma concentration-time curve at steady state (AUCss) of BH-30643 for multiple doses (Phase 1) at steady state. | Predose and up to 24 hours postdose.
  Determine area under the plasma concentration-time curve at steady state (AUCss) of BH-30643.
Objective Response Rate (ORR) | From enrollment until the date of the first documented progression or death from any cause, whichever occurs first, assessed up to study ends or patient discontinue from the study, whichever occurs first (up to approximately 4 years).
  The ORR is defined as a complete response (CR) or partial response (PR) per RECIST v1.1 recorded from first treatment until disease progression or start of new anti-cancer therapy. Both CR and PR must be confirmed by repeat assessments performed no less than 4 weeks after the criteria for response are first met.
Disease Control Rate (DCR) | From enrollment until the date of the first documented progression or death from any cause, whichever occurs first, assessed up to study ends or patient discontinue from the study, whichever occurs first (up to approximately 4 years).
  The DCR is defined as the percentage of subjects whose therapeutic intervention has led to a CR, PR, or stable disease (SD).
Clinical benefit Rate (CBR) | From enrollment until the date of the first documented progression or death from any cause, whichever occurs first, assessed up to study ends or patient discontinue from the study, whichever occurs first (up to approximately 4 years).
  The CBR is defined as the percentage of subjects who achieve a CR, PR, or at least 12 weeks of SD as a result of therapy.
Time to Tumor Response (TTR) | From first dose to the first occurrence of response, assessed up to the date of first documented progression or death from any cause, whichever occurs first (up to approximately 4 years).
  Time to tumor response (TTR) is defined for subjects with a confirmed objective response, as the time from the date of first treatment to the first documentation of objective response (CR or PR) which is subsequently confirmed.
Duration of Response (DOR) | From first occurrence of response until the date of the first documented progression or death from any cause, whichever occurs first, assessed up to study ends or patient discontinue from the study, whichever occurs first (up to approximately 4 years).
  The DOR is defined, for subjects with an objective response per RECIST v1.1, as the time from the first documentation of objective tumor response (CR or PR) to the first documentation of objective tumor progression or death due to any cause, whichever occurs first.
Progression-free Survival (PFS) | From enrollment until the date of the first documented progression or death from any cause, whichever occurs first, assessed up to study ends or patient discontinue from the study, whichever occurs first (up to approximately 4 years).
  The endpoint PFS is defined as the time from the date of the first treatment to the date of the first documentation of objective progression of disease or death due to any cause, whichever occurs first.
Overall Survival | From enrollment until the date of death from any cause, assessed up to study ends or patient discontinue from the study, whichever occurs first (up to approximately 4 years).
  Overall survival is defined as the time from the date of first treatment to the date of death due to any cause.
ERTC-QLC-C30 | From enrollment until the end of treatment, up till patient discontinue from treatment due to any reason (up to approximately 4 years).
  Change from Baseline in Patient Reported Outcome European Organization for Research and Treatment Quality of Life Questionnaire (ERTC-QLC-C30) at Treatment Cycle 2 and beyond (in Phase 1 Part 2 and Phase 2).
NSCLC-SAQ | From enrollment until the end of treatment, up till patient discontinue from treatment due to any reason (up to approximately 4 years).
  Change from Baseline in Patient Reported Outcome Non-Small Cell Lung Cancer Symptom Assessment Questionnaire (NSCLC-SAQ) at Treatment Cycle 2 and beyond (in Phase 1 Part 2 and Phase 2).

CONTACTS AND LOCATIONS:
Locations (38):
- United States (21):
  - Mayo Clinic Hospital - Arizona, Phoenix, Arizona
  - The Regents of the University of California - Irvine, CA Campus, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - University of California, Davis Comprehensive Cancer Center, Sacramento, California
  - Stanford University Medical Center, Stanford, California
  - Yale University - Cancer Center, New Haven, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Mayo Clinic - Florida, Jacksonville, Florida
  - Sarah Cancer Research Institution - Florida Cancer Specialist, Lake Mary, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern Medicine - Northwestern Memorial Hospital Galter Pavilion, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Health, Detroit, Michigan
  - Mayo Clinic Hospital - Rochester, MN, Rochester, Minnesota
  - Thomas Jefferson University, Sidney Kimmel Cancer Center, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, LLC, Nashville, Tennessee
  - The University of Texas - M.D. Anderson Cancer Center, Houston, Texas
  - NEXT Virginia, Fairfax, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
- Australia (2):
  - Austin Health, Heidelberg, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
- Canada (2):
  - Cross Cancer Insitute, Edmonton, Alberta
  - Princess Margaret Cancer Centre, Toronto, Ontario
- Hong Kong (2):
  - Prince of Wales Hospital, Shatin, New Territories
  - Queen Mary Hospital, Hong Kong
- Japan (3):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Kindai University Hospital, Osakasayama-shi, Osaka
  - National Cancer Center Hospital, Tsukiji, Tokyo
- Sarawak General Hosital, Kuching, Sarawak, Malaysia
- Singapore (2):
  - National University Hospital, Kent Ridge
  - National Cancer Centre - Singapore, Singapore
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
- Taiwan (3):
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Cancer Center, Taipei
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Undecided